CLINICAL TRIAL: NCT02465411
Title: Long-term Effects of Continuous Glucose Monitoring in Patients With Type 1 Diabetes Treated With Multiple Daily Insulin Injections - Extension of CGMMDI Trial
Brief Title: Long Term CGM Treatment in Patients With Type 1 Diabetes Treated With Insulin Injections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CGMMDI Extension
Record Dates: First submitted 2015-05-26; First posted 2015-06-08 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2016-11

CONDITIONS: Diabetes Mellitus Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Long-term CGM (Experimental): Continuous glucose monitoring with DexCom G4 platina or later generations during 12 months following participation in the CGMMDI trial
  Interventions: Device: Dexcom G4 or later generation

INTERVENTIONS:
Device: Dexcom G4 or later generation — Continuous glucose monitoring with DexCom G4 platina or later generations

SUMMARY:
A keystone in preventing diabetic complications in patients with type 1 diabetes is good glycaemic control. Frequent self-measurements of blood glucose (SMBG) levels have been an essential part of insulin dosing before meals. However, in recent years continuous glucose monitoring (CGM) has become a treatment option to inform the patient when glucose levels may be too high or low.

In some countries, including Sweden, CGM is reimbursed only when combined with continuous subcutaneous insulin infusions (CSII) in patients with very poor glycaemic control or a history of repeated severe hypoglycaemia in adults with type 1 diabetes. This is based on existing clinical trial data showing a beneficial effect on HbA1c when CGM is combined with CSII. However, despite the fact that the majority of adults with type 1 diabetes are treated with multiple daily insulin injections (MDI), studies on the effect of CGM in patients with type 1 diabetes treated with MDI are sparse. Therefore, the investigators initiated the CGMMDI trial, an ongoing, cross-over clinical trial including 161 MDI patients receiving CGM over 6 months, followed by conventional therapy over six months, with a four-month wash-out period in-between treatment. Evaluations include glycaemic control, hypoglycaemia, quality of life, fear of hypoglycaemia, treatment satisfaction, physical activity, and safety.

From a research or regulatory standpoint, long-term data on treatment effects are expected to a greater extent today than in previous years, due to various reasons, e.g., to evaluate any sustained beneficial effects over time, or long-term patient safety. Accordingly, follow-up of treatment in an extension phase after randomized diabetes trials have become more common over time, especially where many novel glucose-lowering treatments are concerned. Therefore, the aim of the current study is to evaluate long-term effects of CGM in patients with type 1 diabetes treated with MDI. Patients who consent in an extension phase over 1 year of the CGMMDI trial will receive CGM, and evaluations will be performed on sustained glycaemic control effects, hypoglycaemia, glycaemic variability, quality of life, fear of hypoglycaemia, treatment satisfaction, physical activity, and safety.

ELIGIBILITY:
Inclusion Criteria:

* Completion of the CGMMDI trial.
* Written informed consent.

Exclusion Criteria:

* Pregnancy, planned pregnancy for the study duration or pregnancy during the last six months
* Severe cognitive dysfunction or other disease, which is adjudicated by a physician as not suitable for inclusion.
* Required continuous use of paracetamol. Paracetamol must not have been used the week before the study and shall not be used during CGM-use because it disturbs the interpretation of blood glucose levels estimated by the Dexcom. However, other pain killers can be used throughout the study duration.
* History of allergic reaction to any of the CGM materials or adhesives in contact with the skin, or to chlorhexidine or alcoholic anti-septic solution.
* Abnormal skin at the anticipated glucose sensor attachment sites (excessive hair, burn, inflammation, infection, rash, and/or tattoo).
* Other investigator-determined criteria making patients unsuitable for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-06; Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
HbA1c in venous sample | 52 weeks or 78 weeks
  For all variables, measurement at the end of this extension of a cross-over study will be compared to the measurement before long-term CGM was initiated.

SECONDARY OUTCOMES:
Mean glucose level measured by CGM during two weeks. | 52 weeks/78 weeks
Mean Amplitude of Glycemic Excursions (MAGE) measured by CGM during two weeks. | 52 weeks/78 weeks
Standard deviation of glucose levels measured by CGM during two weeks. | 52 weeks/78 weeks
Treatment satisfaction: DTSQs scores | 52 weeks/78 weeks
  Diabetes Treatment Satisfaction Questionnaire (Status)
Well being: WHO 5 scores | 52 weeks/78 weeks
  Questionnaire
Hypoglycemia fear: SWE-HFS scores | 52 weeks/78 weeks
  Swedish Hypoglycaemia Fear Scale Questionnaire
Problem areas: SWE-PAID-20 scores | 52 weeks/78 weeks
  Swedish Problem Areas In Diabetes Questionnaire
Physical activity: IPAQ score | 52 weeks/78 weeks
  International Physical Activity Questionnaire
Treatment experience of CGM score | 52 weeks/78 weeks
  Questionnaire developed for this trial
Proportion of time with low glucose levels measured by CGM during two weeks. | 52 weeks/78 weeks
  Below 3.0 mmol/l and below 4.0 mmol/l, respectively.
Proportion of time with high glucose levels measured by CGM during two weeks. | 52 weeks/78 weeks
  Above 10.0 mmol/l and above 13.9 mmol/l, respectively.
Proportion of time with euglycaemic levels measured by CGM during two weeks. | 52 weeks/78 weeks
  5.5-10.0 mmol/l and 3.9-10.0 mmol/l, respectively.
Proportion of patients lowering their HbA1c by 5 mmol/mol (0.5% in DCCT) or more. | 52 weeks/78 weeks
Proportion of patients lowering their HbA1c 10 mmol/mol (1% in DCCT) or more | 52 weeks/78 weeks
Number of self-reported severe hypoglycaemic events per year | 52 weeks/78 weeks
  Defined as unconsciousness due to hypoglycaemia or need for assistance from another person to resolve hypoglycaemia.

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Lind, MD, PhD, Principal Investigator — NU Hospital Group and University of Gothenburg
Locations (15):
- Sweden (15):
  - Alingsås Hospital, Alingsås
  - Angered Hospital, Angered
  - Ängelholm Hospital, Ängelholm
  - Öbackakliniken, Härnösand
  - Helsingborg Hospital, Helsingborg
  - Central Hospital Kristianstad, Kristianstad
  - Halland Hospital Kungsbacka, Kungsbacka
  - Skåne University Hospital Malmö, Malmo
  - Hospital in Motala, Motala
  - Vrinnevi Hospital, Norrköping
  - University Hospital Örebro, Örebro
  - Södersjukhuset, Stockholm
  - Hospital Trelleborg, Trelleborg
  - NU Hospital Group, Uddevalla
  - Academic Hospital Uppsala, Uppsala

REFERENCES:
- [Derived] Lind M, Olafsdottir AF, Hirsch IB, Bolinder J, Dahlqvist S, Pivodic A, Hellman J, Wijkman M, Schwarcz E, Albrektsson H, Heise T, Polonsky W. Sustained Intensive Treatment and Long-term Effects on HbA1c Reduction (SILVER Study) by CGM in People With Type 1 Diabetes Treated With MDI. Diabetes Care. 2021 Jan;44(1):141-149. doi: 10.2337/dc20-1468. Epub 2020 Nov 15. PMID 33199470